CLINICAL TRIAL: NCT00169273
Title: Epidemiology and Care of Comorbid Obesity and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Minnesota (Other); Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R202009; R01MH068127 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Depression
Keywords: Obesity; Depression; Behavioral; Cognitive; Treatment
MeSH Terms: conditions — Obesity; Depression; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight loss only intervention (Active Comparator): Structured group weight loss intervention
  Interventions: Behavioral: Structured behavioral weight loss group
- Combined intervention (Experimental): Structured group program for weight loss and depression
  Interventions: Behavioral: Weight loss and cognitive-behavioral depression group

INTERVENTIONS:
Behavioral: Structured behavioral weight loss group — Structured group weight loss program
  Arms: Weight loss only intervention
Behavioral: Weight loss and cognitive-behavioral depression group — Structured group program for weight loss and depression
  Arms: Combined intervention

SUMMARY:
We propose to:

* Conduct cross-sectional assessments of depression, disability, health-related quality of life, eating patterns, and eating attitudes in a population-based sample approximately 6000 women aged 40-60 with over-sampling of women with BMI greater than 30 kg/m2.
* Among obese women free of depression, enroll approximately 100 in a 6-month standard behavior therapy weight management program.
* Among obese women with significant depression, randomly assign 200 to either a 6-month standard behavior therapy weight management program or a combined cognitive-behavior therapy program focused on both depression and weight management.
* Complete follow up assessments of weight, depressive symptoms, and functional status in all three treatment groups for 12 months following enrollment

Screening and follow-up data will be used to address the following questions:

* Association between depression and obesity among middle-aged women
* Specific effects of depression and obesity on functional status, disability, and health services utilization
* Impact of depression on participation in and outcomes of a standardized weight management program
* Benefit of combined treatment (focused on depression and weight management) above that of standardized behavioral therapy for obese women with significant depressive symptoms.

DETAILED DESCRIPTION:
Obesity is a significant and growing public health concern, accounting for approximately 300,000 excess deaths per year and approximately 9% of US health care expenditures. Prevalence of obesity has steadily increased, with an estimated rate among middle-aged women exceeding 30%. Obesity has a substantial impact on medical morbidity and health-related quality of life.

Public health approaches to the prevention and treatment of obesity must consider the substantial overlap with depression. Some data suggest a 50% increase in risk of depression among obese women. Women with a history of depression or depression treatment are over-represented among those seeking obesity treatment. Current or past depression is also associated with less success in losing weight or maintaining weight loss. Because women with depressive disorders are typically excluded from clinical trials of weight loss treatments, data on the management of comorbid depression and obesity are limited.

We propose two related studies: A population-based epidemiologic study of the association between obesity and depression among women and a longitudinal study of obesity treatment among two cohorts (one with comorbid obesity and depression, one with obesity only) identified by the epidemiologic study.

Study 1 - Epidemiologic Study: A population-based sample of approximately 6000 women aged 40-65 will complete structured telephone assessment of weight, nutrient intake, physical activity, depression, functional impairment, and disability. Women with Body Mass Index (BMI) >30 will be oversampled. Insurance claims data will be used to measure health care costs. Aims of the epidemiologic study include:

1. Examine the association between obesity and depression among middle-aged women. Secondary analyses will examine possible mechanisms for any association.
2. Examine the specific contributions of obesity and depression to disability, functional impairment, and health care utilization and cost.

Study 2 - Treatment study: A cohort of approximately 100 women with obesity (BMI > 30) and no current depressive disorder will be enrolled in a 6-month state-of-the-art group weight loss treatment. Approximately 200 women with comorbid obesity and depression will be randomly assigned to either the identical weight loss treatment or to a combined cognitive-behavior group therapy program focused on both depression and weight loss. Aims of the treatment study will include:

1. Examine the effect of depression on success in weight loss treatment by comparing weight loss, nutrient intake, and physical activity in depressed and non-depressed women enrolled in the identical weight loss program. Secondary analyses will examine mechanisms for any observed difference.
2. Examine the benefits of a combined weight loss/depression intervention above those of weight loss treatment alone by comparing weight loss, nutrient intake, physical activity, depressive symptoms, functional impairment, and disability in the two groups of women with comorbid obesity and depression randomly assigned to the two different intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 65
* Body Mass Index >= 30
* Clinically significant depression
* PHQ score of 10 or more
* Current or past major depressive episode
* Current symptoms include depressed mood or loss of interest
* Enrolled in Group Health Cooperative health plan

Exclusion Criteria:

* History of treatment for bipolar disorder or schizophrenia
* Not willing to participate in group intervention
* Medical contra-indications to graded exercise program
* Unable to walk for 10 minutes

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2004-04; Primary Completion 2007-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Weight loss since baseline | 24 months
Mean SCL depression score | 24 months

SECONDARY OUTCOMES:
Estimated caloric intake | 24 months
Physical activity | 24 months
Self-efficacy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory E Simon, MD MPH, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Linde JA, Simon GE, Ludman EJ, Ichikawa LE, Operskalski BH, Arterburn D, Rohde P, Finch EA, Jeffery RW. A randomized controlled trial of behavioral weight loss treatment versus combined weight loss/depression treatment among women with comorbid obesity and depression. Ann Behav Med. 2011 Feb;41(1):119-30. doi: 10.1007/s12160-010-9232-2. PMID 20878292